CLINICAL TRIAL: NCT03589131
Title: Robotic-assisted Versus Conventional Laparoscopic Approach for Rectal Cancer Surgery, First Egyptian Academic Center Experience, Randomized Controlled Trial (RCT)
Brief Title: Robotic-assisted Versus Conventional Laparoscopic Approach for Rectal Cancer Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Debakey1
Record Dates: First submitted 2018-05-31; First posted 2018-07-17 (Actual); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms

ARMS (2):
- Robotic-assisted Surgery Group (Active Comparator): In this arm the investigators use a robotic system to perform resection of the rectum harboring the tumor trying to do that while being oncologically safe. The robotic system that we use is the da Vinci Si (Intuitive Surgical, Inc.,Sunnyvale,CA) Interventions used are total operative time, margin assessment, conversion rate to open surgery, baseline demographics, preoperative data and postoperative data
  Interventions: Procedure: Total Operative time; Procedure: Margin assessment; Procedure: Conversion rate to open surgery; Procedure: Baseline demographics; Procedure: Preoperative data; Procedure: Postoperative data
- Laparoscopic Surgery Group (Active Comparator): In this arm the investigators use a Laparoscopy system to perform resection of the rectum harboring the tumor trying to do that while being oncologically safe.
  Interventions used are total operative time, margin assessment, conversion rate to open surgery, baseline demographics, preoperative data and postoperative data
  Interventions: Procedure: Total Operative time; Procedure: Margin assessment; Procedure: Conversion rate to open surgery; Procedure: Baseline demographics; Procedure: Preoperative data; Procedure: Postoperative data

INTERVENTIONS:
Procedure: Total Operative time — Investigators compare the preparation time of the procedure in the operating room and the actual operative time
Procedure: Margin assessment — In this intervention investigators measure the proximal, distal and the important circumferential radial margin away from the tumor to determine if this arm is oncologically safe or not.
Procedure: Conversion rate to open surgery — In this interversion investigators try to measure how much is this arm feasible to completely perform the procedure whether robotically or laparoscopically without conversion to open surgery
Procedure: Baseline demographics — These include gender, age, ASA and BMI. All these data are analyzed and compared in both groups
Procedure: Preoperative data — These include distance of the tumor from the anal verge, clinical stage, whether preoperative chemoradiation "CRT", presence of residual tumor after CRT. All were analyzed and compared
Procedure: Postoperative data — These include pathological stage, number of harvested lymph nodes and immediate postoperative outcome within one month (days of return of bowel function, days of hospital stay, complications, if any, like anastomotic leakage, ileus,wound problems and others, rate of reoperation, rate of readmission & 30-days mortality. All were analyzed and compared

SUMMARY:
This is a prospective randomized controlled study that was conducted on patients of both sexes and definite age group at National Cancer Institute-Egypt and with adenocarcinoma of the rectum located within 15 cm from the anal verge. Tumor localization was categorized as the upper rectum (distal border of tumor is from 10 to 15 cm from the anal verge), middle rectum (5 to 10 cm from the anal verge) or lower rectum (less than 5 cm from the anal verge) as measured by colonoscopy and digital rectal examination. Patients were classified into two groups; robotic assisted rectal surgery and conventional laparoscopic rectal surgery.Baseline demographics (gender, age, ASA, BMI), preoperative data (distance of the tumor from the anal verge, clinical stage, whether preoperative chemoradiation (CRT), presence of residual tumor after CRT, intraoperative data (preparation time, actual operative time, estimated blood loss, conversion rate to open surgery), postoperative data (pathological stage, number of harvested lymph nodes, macroscopic completeness of resection in the form of proximal margin, distal margin, circumferential radial margin) and immediate postoperative outcome within one month (days of return of bowel function, days of hospital stay, complications, if any, like anastomotic leakage, ileus,wound problems and others, rate of re-operation, rate of readmission & 30-days mortality) were analyzed and compared.The criteria for patients selection were the following: histological diagnosis of adenocarcinoma of rectum, no anesthesiological contraindications to minimally invasive surgery, age ≤ 75 years, American Society of Anesthesiologists (ASA) ≤ 2 & the procedures performed by the same surgical team. Patients with metastatic disease, malignant bowel obstruction and those with irresectable tumor were excluded from our study.Preoperative workup (endoscopy with biopsies, radiological imaging including pelvic MRI, liver ultrasound, chest X-ray and routine abdominal and digital rectal examinations) was routinely carried out. The assignment of patients to either group was done by a permuted block randomization. It was an open-labeled study. The study was approved by the institutional review board of National Cancer Institute-Cairo University. All patients provided written informed consent.

DETAILED DESCRIPTION:
Undoubtedly, robotic systems have largely penetrated the surgical field.For any new operative approach to become an accepted alternative to conventional methods, it must be proved safe and result in comparable outcomes. The purpose of this study is to compare the short-term operative as well as oncologic outcomes of robotic assisted and laparoscopic rectal cancer resection.

This is a prospective randomized controlled study that was conducted on all patients of both sexes and definite age group attending the National Cancer Institute and with adenocarcinoma of the rectum located within 15 cm from the anal verge who were eligible to be included in the study. Tumor localization was categorized as the upper rectum (distal border of tumor is from 10 to 15 cm from the anal verge), middle rectum (5 to 10 cm from the anal verge) or lower rectum (less than 5 cm from the anal verge) as measured by colonoscopy and digital rectal examination. Patients were classified into two groups; robotic assisted rectal surgery "The robotic system that we use is the da Vinci Si(Intuitive Surgical, Inc.,Sunnyvale,CA)" and conventional laparoscopic rectal surgery. Baseline demographics (gender, age, ASA, BMI), preoperative data (distance of the tumor from the anal verge, clinical stage, whether preoperative chemo-radiation "CRT", presence of residual tumor after CRT), intraoperative data (preparation time, actual operative time, estimated blood loss, conversion rate to open surgery), postoperative data (pathological stage, number of harvested lymph nodes, macroscopic completeness of resection in the form of proximal margin, distal margin, circumferential radial margin) and immediate postoperative outcome within one month (days of return of bowel function, days of hospital stay, complications, if any, like anastomotic leakage, ileus, wound problems and others, rate of reoperation, rate of readmission & 30-days mortality) were analyzed and compared.The criteria for patients selection were the following: histological diagnosis of adenocarcinoma of rectum, no anesthesiological contraindications to minimally invasive surgery, age ≤ 75 years, ASA ≤ 2 & the procedures performed by the same surgical team. Patients with metastatic disease, malignant bowel obstruction (MBO) and those with irresectable tumor were excluded from our study. Preoperative workup (endoscopy with biopsies, radiological imaging including pelvic MRI, liver ultrasound, chest X-ray and routine abdominal and digital rectal examinations) was routinely carried out. The assignment of patients to either group was done by a permuted block randomization. It was an open-labeled study i.e. patients, investigators (surgeons, researchers) and data collectors knew which procedure will be done to which patients. The study was approved by the institutional review board of the National Cancer Institute, Cairo University. All patients provided written informed consent.

ELIGIBILITY:
Inclusion Criteria:

* histological diagnosis of adenocarcinoma of rectum
* no anesthesiological contraindications to minimally invasive surgery
* age 16 -75 years,
* ASA ≤ 2 &
* the procedures performed by the same surgical team.

Exclusion Criteria:

* Patients with metastatic disease,
* malignant bowel obstruction (MBO) and
* those with irresectable tumor

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2015-04-29 (Actual); Primary Completion 2017-01-12 (Actual); Study Completion 2017-01-12 (Actual)

PRIMARY OUTCOMES:
Operative time of robotic-assisted rectal cancer surgery. | 30 days postoperative
  Comparison of operative time in each arm

SECONDARY OUTCOMES:
Accurate safety margin | 30 days postoperative
  the surgical margins are considered adequate if the proximal, distal and circumferential radial margins are at least 5 cm, 2 cm and 0.1 cm respectively

CONTACTS AND LOCATIONS:
Overall Officials: Yasser A Debakey, Msc, Principal Investigator — Assistant Teacher of Surgical Oncology, National Cancer Institute, Cairo University,Egypt.

IPD SHARING:
Plan to Share IPD: Undecided